CLINICAL TRIAL: NCT02586922
Title: Fetal Lung Volume and Pulmonary Artery Resistance Index Measurement in Term Diabetic Pregnancy and Their Correlation With Neonatal Outcome: a Pilot Study
Brief Title: Fetal Lung Volume and Pulmonary Artery Resistance Index Measurement in Term Diabetic Pregnancy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, Professor Mohamed Laban, Ain Shams University
Other Study IDs: LVPT
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Three-dimensional (3D) ultrasonography — A longitudinal section of fetal chest will be obtained that clearly depicts the lung. A 3D window will be activated . After complete electronic sweep and assurance of absence of fetal or maternal movements to avoid motion artifacts, 3D multi-planar view will be then obtained

SUMMARY:
The aim of this study is to determine cut-off values for fetal lung volume by VOCAL and pulmonary artery resistance index by pulsed Doppler in fetuses of diabetic mothers, and correlate the results with postnatal respiratory distress of the term neonates.

DETAILED DESCRIPTION:
Research question:

Can the assessment of fetal lung volume by Virtual Organ Computed-aided Analysis (VOCAL) and pulmonary artery resistance index by pulsed Doppler predict neonatal respiratory distress syndrome in term fetuses of diabetic mothers?

Research hypothesis:

The assessment of fetal lung volume by VOCAL and pulmonary artery resistance index by pulsed Doppler can predict neonatal respiratory distress syndrome in term fetuses of diabetic mothers.

ELIGIBILITY:
Inclusion Criteria:

-Diabetic pregnant women 38 weeks gestation admitted for elective termination due to various obstetric indications

Exclusion Criteria:

1. Twins.
2. Pregnancy complicated by medical disorders other than Diabetes Mellitus (hypertension, pre-eclampsia, cardiac disorders, thyroid disorders, anemia with pregnancy...etc).
3. Autoimmune disorders.
4. Congenital fetal anomalies.
5. Macrosomia and intrauterine growth restriction (IUGR).
6. Intrauterine fetal death (IUFD).
7. Amniotic fluid index <5cm or >20cm.
8. Patients taking steroids within one week of measurement of lung volume.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a prospective observational study which will be carried out at Ain Shams University Maternity Hospital, Obstetrics and Gynecology department, Faculty of Medicine, Ain Shams University, from December 2015 to December 2016.
  Diabetic pregnant women 38 weeks gestation admitted for elective termination by Caesarian section due to various obstetric indications
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
neonatal respiratory distress | immediately after delivery
  Occurrence of neonatal respiratory distress immediately after delivery utilizing APGAR score at birth in numbers

SECONDARY OUTCOMES:
• Neonatal mortality rate | One week after delivery
  - Follow up for early neonatal mortality rate after Neonatal Intensive Care Unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Laban, Professor, Principal Investigator — Ain Shams University